CLINICAL TRIAL: NCT02809599
Title: Partnered Implementation of Evidence Based Best Care Practice for Benign Paroxysmal Positional Vertigo: A Stepped Wedge, Randomized Controlled Clinical Trial
Brief Title: Evidence Based Best Care Practice for Benign Paroxysmal Positional Vertigo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, William J Meurer, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00109306; R01DC012760 (NIH)
Record Dates: First submitted 2016-06-16; First posted 2016-06-22 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Benign Paroxysmal Positional Vertigo
Keywords: vertigo; dizziness
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Vertigo; Dizziness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-intervention (No Intervention): Patients in hospitals that have not received the intervention (DIZZTINCT) and that meet eligibility criteria will have their medical charts abstracted to assess BPPV processes at the ED Index visit. A random sample of these patients will be contacted by phone for a brief phone interview regarding their recent visit to the Emergency Department for dizziness.
- Post-intervention (Experimental): Patients in hospitals that have received the intervention (DIZZTINCT) and that meet eligibility criteria will have their medical charts abstracted to assess the main study outcome, behavior change in medical providers. A random sample of these patients will be contacted by phone for a brief phone interview regarding their recent visit to the Emergency Department for dizziness.
  Interventions: Behavioral: DIZZTINCT

INTERVENTIONS:
Behavioral: DIZZTINCT — The intervention, DIZZTINCT, is a multi-faceted educational and care-process based intervention designed to improve the guideline-concordant care of patients with BPPV in the emergency department. The intervention includes six main components: the recruitment and training of local champions who will serve as colleague experts in the community; interactive hands-on educational sessions that address BPPV mechanisms, evidence and practice; a high-yield decision-aid web application for self study and point of care use; development of a referral network for follow up care; follow-up educational sessions to review successes and barriers amongst the intervention group; and other resources developed locally in partnership with the community medical providers.
  Arms: Post-intervention

SUMMARY:
The study evaluates a theory-based educational intervention and implementation strategy on the use of the Dix-Hallpike test (DHT) and Canalith Repositioning Maneuver (CRM) in a community Emergency Department (ED) setting. The DHT and CRM are used to diagnose and treat Benign Paroxysmal Positional Vertigo (BPPV).

DETAILED DESCRIPTION:
The Dix-Hallpike Test (DHT) and Canalith Repositioning Maneuver (CRM) are used to diagnose and treat Benign Paroxysmal Positional Vertigo (BPPV). BPPV processes have an evidence base that is at the clinical practice guideline level. The DHT is the gold standard test for DHT and the CRM is supported by numerous randomized controlled trials and systematic reviews.

The problem is that BPPV processes are substantially underutilized.

This study looks to increase the use of BPPV processes within a community ED setting by implementing a theory-based educational intervention. The unit of randomization and target of intervention is the hospital. After an initial observation period, the six community hospitals will undergo the intervention in five waves (the smallest two hospitals will be paired). The order will be randomized. This is a partnered research project with local physicians engaging in best practice implementation.

Sample Size

The trial will start with an initial no intervention period of approximately 4 months followed by randomized staggered intervention with a new hospital entering approximately every 2 months, finalized by approximately 4 post-intervention months will result in the approximately balanced number of 867 visits occurring without intervention and 933 visits occurring under (post) intervention. This calculation assumes the average anticipated total patient visit rate of 100 patients per month. Based on our pilot studies and the literature we expect the DHT or CRM procedure to be done in 5% patients before the intervention. With the expected number of visits calculated above, we will be able to detect the increased DHT or CRM rate of 9% and above with 90% power by a two-sided test at the significance level of 5%. We expect a much bigger difference of 5% vs. 20% pre- vs. post-intervention DHT/CRM rates, respectively. Under this expected difference, we will have the power exceeding 99%. In fact, an order of magnitude smaller visit rate of 10.4 patients per month would be sufficient for 90% power under the anticipated difference. The reserves of power will be used to provide more power to fine-tune the multivariate mixed regression models and associated secondary analyses.

Data Analyses

The intervention is delivered to hospitals. Intervention is a binary variable with two levels, pre-intervention (no intervention), post-intervention (under intervention).

The primary analysis will use binary logistic regression and will include covariates for hospital, month (to handle secular trends), and intervention (see below). For a set of new patient visits, the binary random variable DHT/CRM/referral yes/no will serve as the primary response. Patient visits will be supplied with patient-, hospital- and provider-level covariates as well as the calendar time variable modeling the secular trend, and the intervention yes/no variable measuring whether the visit occurs under intervention or not. To take hospital- and provider-specific unmeasured features into account, hospital and provider categorical variables will be included in the analysis. Due to the fact that the number of hospitals and providers is much smaller than the number of patient visits, adjusting for hospital and provider effects by way of categorical variables will not lead to bias. Secondary analyses will explore alternative approaches using random effects (Gaussian) models. A two-sided model-based test for the intervention variable will be used to test the primary hypothesis at the significance level of 5%.

The secondary analysis (safety) will numerically summarize the 90-day stroke rate - cumulatively and stratified for stroke diagnosed on the index dizziness visits and for post index visit strokes (delayed diagnosis) in patients seen at EDs with and without the intervention. This is anticipated to be very rare. The intervention does not target improving stroke diagnosis. However, evaluating both the index visit stroke diagnosis rate and the delayed diagnosis rate should allow for determination of major changes. We anticipate the index visit stroke diagnosis rate to be approximately 2% and the delayed diagnosis rate approximately to be 1%.

ELIGIBILITY:
Inclusion Criteria:

* ED patient seen at one of six full service non-freestanding Emergency Departments in Nueces County, Texas
* Principal dizziness case: the triage reason for visit is a dizziness symptom OR a dizziness symptom is one of first three listed complaints in physician medical record OR a dizziness diagnosis (e.g., dizziness or vertigo NOS, BPPV, vestibular neuritis) is recorded as one of the first three final ED diagnoses.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7635 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2018-04-14 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
Likelihood of Receiving a BPPV Care Process | Index ED Visit (within hours to 2 days)
  Pre-intervention (no intervention) vs. post-intervention (under intervention).The primary endpoint is measured at the individual patient level, and is the presence of documentation of either the Dix-Hallpike test, the Epley Maneuver (or CRM) (since the first step of the CRM is the diagnostic maneuver).

SECONDARY OUTCOMES:
Outpatient Referral to a BPPV Provider | Index ED Visit (within hours to 2 days)
  Pre-intervention (no intervention) vs. post-intervention (under intervention) rate of referral to a BPPV provider
90-day Cumulative Incidence of Stroke | 90 days following initial ED discharge home visit for dizziness
  Stroke diagnosed on the index dizziness visits and for post index visit strokes (delayed diagnosis) within the dizziness population aged 45 and older seen in EDs that have received the intervention versus patients seen in EDs that have not received the intervention.

OTHER OUTCOMES:
Stroke at Index ED Dizziness Visit | Index ED Visit (within hours to 2 days)
ED Length of Stay | Index ED Visit (within hours to 2 days)
Neuroimaging utilization | Index ED Visit (within hours to 2 days)
  Was CT, MRI, or vascular imaging performed in the ED
Inpatient hospitalization Utilization | Index ED Visit (within hours to 2 days)
  Was the patient admitted to the hospital from the ED

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Kerber, MD, Principal Investigator — University of Michigan; William Meurer, MD, Principal Investigator — University of Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kerber KA, Damschroder L, McLaughlin T, Brown DL, Burke JF, Telian SA, Tsodikov A, Fagerlin A, An LC, Morgenstern LB, Forman J, Vijan S, Rowell B, Meurer WJ. Implementation of Evidence-Based Practice for Benign Paroxysmal Positional Vertigo in the Emergency Department: A Stepped-Wedge Randomized Trial. Ann Emerg Med. 2020 Apr;75(4):459-470. doi: 10.1016/j.annemergmed.2019.09.017. Epub 2019 Dec 20. PMID 31866170
- [Derived] Meurer WJ, Beck KE, Rowell B, Brown D, Tsodikov A, Fagerlin A, Telian SA, Damschroder L, An LC, Morgenstern LB, Ujhely M, Loudermilk L, Vijan S, Kerber KA. Implementation of evidence-based practice for benign paroxysmal positional vertigo: DIZZTINCT- A study protocol for an exploratory stepped-wedge randomized trial. Trials. 2018 Dec 22;19(1):697. doi: 10.1186/s13063-018-3099-0. PMID 30577834